CLINICAL TRIAL: NCT07207473
Title: Helping Veterans With Obstructive Sleep Apnea Determine What Matters Most in Choosing a Treatment Option: a Randomized Trial
Brief Title: Behavioral Optimization to Overcome Obstructive Sleep Apnea Treatment Barriers
Acronym: BOOST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PULM-005-25S
Record Dates: First submitted 2025-09-26; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Sleep Apnea
Keywords: sleep apnea; decision making, shared; health priorities
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep education program X + Y (Experimental): Brief 4 session education program with sleep specialist focused on behavioral strategies for improving use of sleep apnea therapy. Tests behavioral strategy program X plus Y.
  Interventions: Behavioral: Behavioral strategy program X plus Y
- Sleep education program X (Active Comparator): Brief 4 session education program with sleep specialist focused on behavioral strategies for improving use of sleep apnea therapy Tests behavioral strategy X.
  Interventions: Behavioral: Behavioral strategy program X

INTERVENTIONS:
Behavioral: Behavioral strategy program X plus Y — Brief 4 session education program with sleep specialist focused on behavioral strategies for improving use of sleep apnea therapy. Tests behavioral strategy program X plus Y.
  Arms: Sleep education program X + Y
Behavioral: Behavioral strategy program X — Brief 4 session education program with sleep specialist focused on behavioral strategies for improving use of sleep apnea therapy Tests behavioral strategy X.
  Arms: Sleep education program X

SUMMARY:
Previous studies have shown that programs encouraging the use of OSA treatments can help patients use these treatments more often, but the improvement is usually modest. This trial will test if giving patients a decision-making tool when they are first diagnosed with OSA, and combining their responses from this tool into a supportive program, will improve sleep quality and help them use their treatment more regularly.

DETAILED DESCRIPTION:
Background and Significance:

Obstructive Sleep Apnea (OSA) is a significant health issue for many middle-aged and older Veterans. This condition can lead to daytime sleepiness and poor sleep quality and is a risk factor for more serious conditions such as cardiovascular disease, cognitive decline, and even increased risk of death. Common treatments for OSA include the use of medical devices such as positive airway pressure machines or oral appliances. However, many Veterans find these devices uncomfortable or difficult to use regularly. This clinical trial aims to test a new 4 session program to help Veterans stick to their OSA treatment plans using a more person-centered approach.

Innovation and Impact:

This innovative, person-centered approach is integral to the VA's "age-friendly" healthcare transformation. By focusing on what matters most to older Veterans, the investigators aim to enhance their compliance with, and the effectiveness of, OSA therapy. Aligning OSA treatment decisions with each Veteran's health priorities is expected to improve their overall wellbeing and make OSA treatments more effective.

Specific Aims:

1. Improve Sleep Quality: To determine if the new program improves patient-reported outcomes, specifically sleep quality.
2. Enhance Therapy Adherence: To evaluate if the new program increases acceptance and adherence to OSA device therapy.
3. Align Treatment with Priorities: To assess the impact of the program on ensuring that treatment decisions align with each patient's health priorities and values.

Methodology: The investigators will conduct a 5-year multi-site randomized controlled trial with a total of 128 Veterans across sites, aged 50 and older who have been newly diagnosed with OSA. Participants will be randomly assigned to either the new program or an active-control program (both programs include 1 self-directed session and 3 sessions delivered by sleep providers) that incorporate behavioral adherence strategies currently used in the investigators sleep centers. The research team will measure the outcomes 6 months after the program ends.

Path to Translation/Implementation:

The long-term goal of this work is to improve sleep quality and use of prescribed OSA therapies among middle-aged and older Veterans with OSA. If successful, the investigators will implement the intervention at the investigators' institutions and conduct a future type 2 hybrid design trial to test both the effectiveness of the program and its potential for wider implementation.

ELIGIBILITY:
Inclusion Criteria:

* referred for an overnight diagnostic sleep test to evaluate for sleep-disordered breathing during the study period
* currently untreated for OSA (not prescribed therapy in the past year)

Exclusion Criteria:

* referral for overnight sleep test is for another reason than to diagnosis sleep-disordered breathing
* unable to read printed material (e.g., magazine) in English language
* unable to write
* unstable medical/psychiatric illness (e.g., recent hospitalization)
* Telephone Mini-Mental State Examination (MMSE) < 21 or diagnosis of dementia
* unstable housing
* unable to attend study video or in-person visits

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 6-months after the end of the intervention/control sessions, which is approximately 8 months after randomization.
  The PSQI total score will be used as a measurement of sleep quality. Scores range from 0 to 21. Higher scores indicate worse outcome.

SECONDARY OUTCOMES:
Acceptance of therapy | One week after the end of the intervention/control sessions, which is approximately 2 months after randomization.
  Percentage of participants prescribed device therapy with > 0 days of use in the 30 days prior to the 6-month follow-up timepoint.
Treatment adherence by machine report | 6-months after the end of the intervention/control sessions, which is approximately 8 months after randomization.
  Percentage of days of machine reported use >= 4 hours in the prior 30 days.

OTHER OUTCOMES:
Decisional Conflict Scale - 1 item | End of session 1, which is within 7 days of randomization.
  Decisional Conflict Scale "What's important" item. This item is scored as 0 (best) to 4 (worst).

CONTACTS AND LOCATIONS:
Overall Officials: Constance H Fung, MD MSHS, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (2):
- United States (2):
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No